CLINICAL TRIAL: NCT00151502
Title: An 80-Week, Randomized, Multi-Center, Parallel-Group, Double-Blind Study of the Efficacy and Safety of Atorvastatin 80 MG Plus an Acetylcholinesterase Inhibitor Versus an Acetylcholinesterase Inhibitor Alone in the Treatment of Mild to Moderate Alzheimer's Disease.
Brief Title: To Evaluate the Safety and Effectiveness of Atorvastatin Plus a Cholinesterase Inhibitor in AD Patients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A2581078
Record Dates: First submitted 2005-09-06; First posted 2005-09-09 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin

SUMMARY:
The purpose of this study is to find out if atovastatin, when taken with a cholinesterase inhibitor, is effective for treating Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic evidence of probable Alzheimer's disease consistent with NINCDS/ADRDA and DSM IV criteria.
* Subject's Mini-Mental Status Examination Score (MMSE) must be in the range of 13 - 25 (inclusive) at Screening.

Exclusion Criteria:

* Subjects with dementia due to causes other than Alzheimer's disease.
* Any condition, which, in the investigator's judgment might increase the risk to the subject or decrease the reliability of the data required to meet the objectives of the study.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2002-11; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
If the results of this study demonstrate efficacy and lead to the approval by the FDA of atorvastatin for use in humans for the treatment of Alzheimer's disease, this would be available as an additional treatment option for patients.

SECONDARY OUTCOMES:
If the results of this study demonstrate efficacy and lead to the approval by the Food and Drug Administration of atorvastatin for use in humans, subject activities of daily living are being assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (90):
- United States (38):
  - Pfizer Investigational Site, Sun City, Arizona
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, Laguna Hills, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Fort Lauderdale, Florida
  - Pfizer Investigational Site, Fort Myers, Florida
  - Pfizer Investigational Site, Miami Beach, Florida
  - Pfizer Investigational Site, Pompano Beach, Florida
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Fort Wayne, Indiana
  - Pfizer Investigational Site, Paducah, Kentucky
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, South Dartmouth, Massachusetts
  - Pfizer Investigational Site, West Yarmouth, Massachusetts
  - Pfizer Investigational Site, Worcester, Massachusetts
  - Pfizer Investigational Site, Kalamazoo, Michigan
  - Pfizer Investigational Site, Jamesburg, New Jersey
  - Pfizer Investigational Site, Princeton, New Jersey
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Troy, New York
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Allentown, Pennsylvania
  - Pfizer Investigational Site, Jenkintown, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, East Providence, Rhode Island
  - Pfizer Investigational Site, Providence, Rhode Island
  - Pfizer Investigational Site, Madison, Tennessee
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Wichita Falls, Texas
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Madison, Wisconsin
  - Pfizer Investigational Site, Milwaukee, Wisconsin
- Australia (7):
  - Pfizer Investigational Site, East Gosford, New South Wales
  - Pfizer Investigational Site, Randwick, New South Wales
  - Pfizer Investigational Site, Daw Park, South Australia
  - Pfizer Investigational Site, Woodville South, South Australia
  - Pfizer Investigational Site, Ballarat, Victoria
  - Pfizer Investigational Site, WEST Heidelberg, Victoria
  - Pfizer Investigational Site, Nedlands, Western Australia
- Austria (2):
  - Pfizer Investigational Site, Vienna
  - Pfizer Investigational Site, Wein
- Canada (8):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Québec, Quebec
  - Pfizer Investigational Site, Verdun, Quebec
- Denmark (5):
  - Pfizer Investigational Site, Aarhus
  - Pfizer Investigational Site, Copenhagen
  - Pfizer Investigational Site, Hillerød
  - Pfizer Investigational Site, Rudkøbing
  - Pfizer Investigational Site, Svendborg
- Germany (8):
  - Pfizer Investigational Site, Bad Honnef
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Bochum
  - Pfizer Investigational Site, Bonn
  - Pfizer Investigational Site, Göttingen
  - Pfizer Investigational Site, Hanover
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Tübingen
- South Africa (5):
  - Pfizer Investigational Site, Rosebank, Gauteng
  - Pfizer Investigational Site, Willows, Gauteng
  - Pfizer Investigational Site, Pinetown, KwaZulu-Natal
  - Pfizer Investigational Site, Belleville
  - Pfizer Investigational Site, Westville
- Spain (3):
  - Pfizer Investigational Site, Terrassa, Barcelona
  - Pfizer Investigational Site, Barcelona
  - Pfizer Investigational Site, Madrid
- Sweden (5):
  - Pfizer Investigational Site, Linköping
  - Pfizer Investigational Site, Malmo
  - Pfizer Investigational Site, Mölndal
  - Pfizer Investigational Site, Stockholm
  - Pfizer Investigational Site, Uddevalla
- United Kingdom (9):
  - Pfizer Investigational Site, Bradford, England
  - Pfizer Investigational Site, Stirling, Stirlingshire
  - Pfizer Investigational Site, Swindon, Wiltshire
  - Pfizer Investigational Site, Bath
  - Pfizer Investigational Site, Belfast
  - Pfizer Investigational Site, Glasgow
  - Pfizer Investigational Site, Penarth
  - Pfizer Investigational Site, Southhampton
  - Pfizer Investigational Site, Stirling

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2581078&StudyName=To%20Evaluate%20the%20Safety%20and%20Effectiveness%20of%20Atorvastatin%20Plus%20a%20Cholinesterase%20Inhibitor%20in%20AD%20Patients.